CLINICAL TRIAL: NCT07051317
Title: Establishment and Application Evaluation of a Precise and Accurate Measurement Method for Retinal Hemodynamics Based on Adaptive Optics Scanning Laser Ophthalmoscopy (AOSLO)
Brief Title: AOSLO-Based Precise Measurement of Retinal Hemodynamics: Development and Application Assessment
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KYPJ100
Record Dates: First submitted 2025-06-18; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-02

CONDITIONS: Myopia, High-Grade; Myopia; Refractive Error
Keywords: Myopia, High-Grade; Adaptive optics; Retinal hemodynamics
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myopia, low and middle grade
- myopia, high grade

SUMMARY:
Changes in retinal hemodynamics play a key role in the development of various eye diseases. Currently, mainstream hemodynamic evaluation techniques have low resolution and poor measurement accuracy, limiting their widespread application. Adaptive optical laser scanning ophthalmoscopy (AO-SLO) can capture retinal vascular images at the cellular level, offering the potential for high-precision retinal hemodynamic evaluation. This project will: ① innovate the AO-SLO blood flow imaging scanning module and acquisition mode, develop algorithms for extracting spatiotemporal signal features from blood flow images, and achieve quantitative analysis of retinal hemodynamics based on AO-SLO; ② construct an in vitro retinal hemodynamic measurement simulation eye, conduct multidimensional AO-SLO hemodynamic measurements, and establish an intelligent model for precise calibration of retinal hemodynamic parameters; ③ conduct AO-SLO-based retinal hemodynamic studies in high myopia, integrating multi-modal ophthalmic imaging to investigate the patterns of changes in retinal vascular structure and blood flow function in high myopia. Ultimately, a new precision measurement imaging technology platform for retinal hemodynamics will be established.

DETAILED DESCRIPTION:
The retina is the initial site where the eye receives external light and forms vision, and it is also the site where various blinding eye diseases occur. Retinal diseases such as diabetic retinopathy (DR), high myopia-related retinal disease, and age-related macular degeneration (AMD) impose a significant visual burden worldwide. The retinal vascular system is involved in the nutrient supply and waste transport of retinal cells, and the integrity of its structure and function is the foundation for maintaining retinal function. Therefore, assessing changes in retinal blood flow can help understand the mechanisms underlying disease progression, thereby promoting early diagnosis and precise treatment of retinal diseases.

Retinal vessels are the only circulatory system in the human body that can be directly observed, allowing for direct visualization and assessment of changes in hemodynamic characteristics such as retinal vascular blood flow velocity. Traditional fluorescein fundus angiography (FFA) involves intravenous injection of fluorescein to indirectly assess retinal perfusion velocity by observing the distribution of fluorescein in the retinal vascular system over time. However, FFA is an invasive procedure and is not suitable for evaluating early hemodynamic changes.

With the development of ophthalmic imaging technology, new fundus imaging techniques can provide more objective, convenient, and non-invasive tools for measuring blood flow velocity. Currently, mainstream hemodynamic evaluation devices, such as laser Doppler, retinal function imaging (RFI), and laser speckle technology, can quantify parameters such as blood flow velocity, blood flow volume, and vascular resistance by extracting spatiotemporal imaging signals of red blood cell movement or analyzing the optical effects caused by movement. However, these devices are limited in clinical application due to issues such as low resolution, low measurement accuracy, and poor reproducibility.

Adaptive optics (AO) is a technology that corrects aberrations and improves the imaging resolution of optical systems. By combining high-definition fundus scanning with a scanning laser ophthalmoscope (SLO), it is possible to achieve cellular-level resolution imaging and quantitative analysis of retinal vascular structures. By using AO-SLO to collect high spatio-temporal resolution image sequences of retinal vessels, it is possible to establish a novel method for evaluating retinal hemodynamics, enabling precise and stable measurements of blood flow velocity and blood flow volume.

Myopia is a highly prevalent eye disease worldwide, with an estimated prevalence exceeding 50% by 2050. Compared to moderate and low myopia, high myopia significantly increases the incidence of macular degeneration and glaucoma. The exact mechanisms underlying the pathological changes in high myopia remain controversial, but increasing evidence suggests that blood flow alterations may be a key pathological mechanism in high myopia-related retinal diseases. Due to the lack of objective evaluation methods, the patterns of hemodynamic changes in high myopia remain unclear. In summary, there is currently a lack of objective, precise hemodynamic quantification assessment tools in ophthalmic clinical practice. Developing a novel retinal hemodynamic imaging assessment model based on AO-SLO, establishing precise hemodynamic measurement methods, and achieving real-time, non-invasive, high-resolution imaging and quantitative analysis of retinal blood flow in living human eyes will provide important imaging evidence for the early diagnosis of retinal diseases such as high myopia-related retinal lesions.

This project will Innovate the AO-SLO blood flow imaging scanning module and acquisition mode, develop algorithms for extracting spatio-temporal signal features from blood flow images, and achieve quantitative analysis of retinal hemodynamics based on AO-SLO; construct an in vitro retinal hemodynamic measurement simulation eye, conduct multi-dimensional AO-SLO hemodynamic measurements, and establish an intelligent model for precise calibration of retinal hemodynamic parameters; conduct AO-SLO-based retinal hemodynamic studies in high myopia, integrating multi-modal ophthalmic imaging to investigate the patterns of changes in retinal vascular structure and blood flow function in high myopia. Ultimately, a new precision measurement imaging technology platform for retinal hemodynamics will be established.

This study will analyze the following indicators: retinal blood flow velocity, flow velocity standard deviation, flow rate, vessel diameter, lumen diameter, wall thickness, wall-to-lumen ratio, vascular density, diameter, and tortuosity measurements in participants with high myopia and non-high myopia one week after enrollment. Quantitative data will be described using mean ± standard deviation (M±SD), and differences between the two groups will be analyzed, along with correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must understand the clinical study and voluntarily participate, and sign an informed consent form;
2. Age 18-30 years old, no gender restrictions;
3. Equivalent spherical power≤0D cylindrical power -2.0D to +2.0D, best-corrected visual acuity ≥ 1.0

Exclusion Criteria:

1. Participants with significant refractive media opacity-related conditions (severe cataracts, vitreous diseases, corneal diseases, etc.) at screening, or unable to complete or cooperate with routine ophthalmic examinations;
2. History of or concurrent conditions such as ptosis, nystagmus, diabetic retinopathy, various macular degeneration, retinal vascular diseases, optic nerve inflammatory diseases, primary angle-closure glaucoma, various secondary glaucoma, amblyopia, or severe strabismus
3. History of previous eye surgery
4. Patients with severe hypertension, diabetes, or other systemic diseases that cause secondary changes in the retina
5. Patients with posterior scleral staphyloma, lacquer cracks, choroidal neovascularization, or Fuchs' spots
6. Pregnant women, breastfeeding women, monocular individuals, and individuals with disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The people From Guangzhou, Guangdong Province, China
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood flow velocity in the central arteries and veins of the retina | 7 days after the enrollment
  Measure the blood flow velocity and flow velocity standard deviation of the central arteries and veins of the retina of the subject using an adaptive optical laser scanning ophthalmoscope.
The structure of central retinal arteries and veins | 7 days after the enrollment
  Measure the diameter of the central arteries and veins of the retina, the thickness of the vessel walls, and the wall-to-lumen ratio of the subjects using an adaptive optics laser scanning ophthalmoscope.
Retinal and choroidal capillary morphological parameters | 7 days after the enrollment
  Use OCTA to obtain images of superficial and deep capillaries and choroidal capillaries within a 3×3 mm area of the posterior pole of the retina, and use a proprietary algorithm to extract morphological parameters.

SECONDARY OUTCOMES:
The examination for anterior segment of eyes | Baseline
  Use a slit lamp microscope to examine the cornea, conjunctiva, anterior chamber, lens, and other anterior structures of the anterior segment of the eye
Axis of the eye | Baseline
  Measure the axial length of the subject's eye using the IOL-Master 500
Best corrected vision cutiy | Baseline
  Assess the best corrected vision by subjective refraction
Intraocular pressure | Baseline
  Measure intraocular pressure in both eyes using a non-contact tonometer.
Fundus color photography | Baseline
  Using non-mydriatic fundus photography to obtain images of the posterior pole of the retina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR